CLINICAL TRIAL: NCT04659473
Title: COVID-19, the Third Wave Update People Coping With the COVID-19. A Cross-sectional Online Spanish Survey
Brief Title: Spanish Survey on Third Wave of COVID-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Beatriz-María Bermejo-Gil, Professor, University of Salamanca
Other Study IDs: CovidSal01/2020
Record Dates: First submitted 2020-12-08; First posted 2020-12-09 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Covid19
Keywords: COVID-19; Epidemiology; Signs and Symptoms; Spain; Rapid online survey
MeSH Terms: conditions — COVID-19; Signs and Symptoms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Online survey — This study aims to apply a rapid online survey to determine the Spanish situation in this third wave of the pandemic.

SUMMARY:
Due to the pandemic situation, a rapid online survey may be the best method to assess and track people's pandemic cooping. Regarding the huge media influence and the government's restrictions to control the spread of covid-19; it is needed to know more about people's perception and situation to conduct future contentions plans. This study aims to apply a rapid online survey to determine the Spanish situation in this third wave of the pandemic. The survey will be delivered to 1000 participants to obtain a representative sample. It would be divided into six sections (general information, demography data, social and consuming habits, Covi-19 question, questions for Covid-19 positive, and questions for Covid-19 negative).

ELIGIBILITY:
Inclusion Criteria:

* Owning online connection
* Ability to answer and complete the survey

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The sample was selected from the Spanish community population
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-09 (Estimated); Primary Completion 2020-12-20 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
What's your work or study system nowadays? | 20 seconds
  Multiple choice questionnaire
Habits before the Covid-19 pandemic | 60 seconds
  Likert scale questionnaire
Habits in the Covid-19 pandemic | 60 seconds
  Likert scale questionnaire
Personal Covid-19 exposure and disease | 10 seconds
  Dichotomous options questionnaire
Positive Covid-19: tests, diagnosis, symptoms and quarantine | 60 seconds
  Multiple choice questionnaire
Negative Covid-19: tests and quarantine | 40 seconds
  Multiple choice questionnaire
Expectations | 10 seconds
  Multiple choice questionnaire

SECONDARY OUTCOMES:
Date of birth | 20 seconds
  It is registered in the survey to know the age
Sex | 20 seconds
  It is registered in the survey
Height | 20 seconds
  It is registered in centimeters
Weight | 20 seconds
  It is registered in kilograms
Blood type | 20 seconds
  Multiple choice questionnaire
Pathologic history | 20 seconds
  Multiple choice questionnaire
Region of residence | 20 seconds
  Multiple choice questionnaire
City of residence | 20 seconds
  Multiple choice questionnaire
Rural or urban environment | 20 seconds
  Dichotomous options questionnaire
Cohabitants in the family unit | 20 seconds
  The number of cohabitants is registered in the survey

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz M Bermejo-Gil, Professor, Principal Investigator — University of Salamanca
Locations (1):
- Universidad de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided